CLINICAL TRIAL: NCT02038816
Title: A PHASE II STUDY OF Azacitidine Plus Deferasirox (ICL670) in Higher Risk Myelodysplastic Syndromes (MDS)
Brief Title: Azacitidine Plus Deferasirox (ICL670) in Higher Risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual too slow, insufficient patients
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ACA02T
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deferasirox + Azacitidine (Experimental): Azacitidine 75 mg/m2 daily X 7 days every 28 days for 6 cycles + Deferasirox 10-30 mg/kg/d depending on transfusion needs
  Interventions: Drug: Deferasirox + Azacitidine; Drug: Azacitidine
- Azacitidine (Active Comparator): Azacitidine 75 mg/m2 daily X 7 days every 28 days for 6 cycles
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Deferasirox + Azacitidine — Deferasirox:
  20 mg/kg/d for < 14ml/kg/mo pRBCs (~ <4U/mo), 30mg/kg/d for ≥14ml/kg/mo pRBCs(≥4U/mo), 10mg/kg/d for transfusion-independent patients
  Other Names: Exjade; Vidaza
  Arms: Deferasirox + Azacitidine
Drug: Azacitidine — Azacitidine 75mg/m2 sc daily X 7 days (5-2-2 schedule permitted) on a 28 day cycle for 6 cycles
  Other Names: Vidaza

SUMMARY:
Myelodysplastic syndromes are common blood disorders that can affect as many as one in 1000 Canadians over the age of 65. They are characterized by low blood counts that require frequent blood transfusions. The development of iron overload in these patients is inevitable. The iron deposits in vital organs such as the heart and the liver and can lead to organ dysfunction. Deferasirox is a well-studied drug that helps remove iron from the body. Most people with this disorder die due to progression of their disease to acute leukemia through multiple mechanisms. Iron overload in patients with myelodysplastic syndromes has been shown to be associated with shorter survival, and potentially a higher chance of leukemia. In a certain sub-group of higher risk patients, the drug azacitidine has been shown to decrease the chance of progression to leukemia and death from it. Thus, it is presently the standard of care for these patients. However, 50% of higher risk patients are still unresponsive to this medication, leaving a large group of patients for which other treatment options are emergently needed. Given that a large proportion of higher risk MDS patients fail to respond to azacitidine, and the evidence that iron deposition may lead to increased leukemic transformation, we would like to study whether iron removal from the body with deferasirox potentiates azacitidine in its effects on overall survival, as well as the chance of leukemia transformation. This question needs to be addressed in a randomized controlled trial, and the first step is a preliminary study to determine if the combination of azacitidine and deferasirox has any biologic effect. This study will determine whether this combination leads to blood count improvement over azacitidine alone. If this drug combination ultimately proves more useful than azacitidine alone with respect to survival, this has the potential to impact the care of a large proportion of patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
Patients with stable disease after 6 cycles of AZA with higher risk MDS will be randomized to either standard of care (continued AZA until progression ) or AZA + defasirox. Primary endpoint is augmented response rate by the addition of deferasirox

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 yrs of age
* WHO defined MDS with Higher risk MDS (IPSS int-2/high)
* Azacitidine X at least 6 cycles with no hematologic improvement/no disease progression as per IWG 2006 criteria
* Ferritin >500 µg/L
* If transfusion independent, must have Hb <110 g/L OR Neutrophils < 1,000/mL OR Platelets < 100,000/mL
* ECOG ≤2
* CrCl >40 ml/min

Exclusion Criteria:

* Increased ALT (>300 U/L)
* Uncontrolled infection
* HIV+
* Pregnant or breast-feeding
* Previous and concurrent iron chelation
* Concurrent use of hematopoietic growth factors including erythropoietin, darbepoietin and granulocyte colony stimulating factor
* Concurrent use of other disease modifying agents including cytotoxic chemotherapy, histone deacetylase inhibitors, other hypomethylating agents or lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of patients with hematologic improvement as defined by the IWG criteria30 with the addition of deferasirox to azacitidine compared with azacitidine alone in higher risk non-responding MDS patients after 6 cycles of azacitidine. | 6 months
  improvement in blood counts or remission status

SECONDARY OUTCOMES:
Tolerability (defined by the percentage of patients able to remain on deferasirox for 6 cycles concurrent with azacitidine) and safety (type, using CTCAE version 4.0, frequency, severity, and relationship of adverse events to study therapy) | 6 months
  toxicity as defined by compliance
Percentage and absolute change in serum ferritin and labile plasma iron (LPI) between baseline and end of study | 6 months
  Impact of experimental arm on iron parameters
Percentage change in CD34 cell intracellular reactive oxygen species (ROS) from baseline to end of study. | 6 months
  Impact of experimental arm on markers of oxidative stress in the bone marrow
Percentage change in erythroid colony forming units (BFU-E and CFU-E) from baseline to end of study | 6 months
  Impact of experimental arm on erythropoiesis
Percentage change in markers of DNA damage (lipid peroxidation, GSH content, and gH2AX expression), and activity of NFkappaB and Akt signaling pathways between baseline and end of study. | 6 months
  Impact of experimental arm on markers of DNA damage

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD, Principal Investigator — Odette Cancer Center
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No